CLINICAL TRIAL: NCT03297788
Title: Whole Brain Radiation Therapy (WBRT) Alone Versus Radiosurgery (SRS) for Patients With 1-10 Brain Metastases From Small Cell Lung Cancer
Brief Title: Whole Brain Radiation Therapy Alone vs. Radiosurgery for SCLC Patients With 1-10 Brain Metastases
Acronym: ENCEPHALON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juergen Debus (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Director of the Department Radiation Oncology, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCEPHALON
Record Dates: First submitted 2017-09-19; First posted 2017-09-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: SCLC; Brain Metastases
Keywords: SCLC; Brain Metastases; SRS (stereotactic radiosurgery); WBRT (whole brain radiotherapy)
MeSH Terms: conditions — Brain Neoplasms; Snyder Robinson syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: SRS (Experimental): Patient receive stereotactic radiosurgery (SRS), dose prescription according to the size of radiated brain metastases
  Interventions: Radiation: SRS
- Arm B: WBRT (Active Comparator): Patients receive whole brain radiotherapy (WBRT)
  Interventions: Radiation: WBRT

INTERVENTIONS:
Radiation: SRS — For SRS the dose prescription to the PTV will be as follows:
  * 20 Gy to the 70%-isodose (lesions < 2 cm max. diameter)
  * 18 Gy to the 70%-isodose (lesions 2 - 3 cm max. diameter)
  * 6 x 5 Gy to the conformally surrounding isodose (lesions > 3 cm max. diameter)
  Arms: Arm A: SRS
Radiation: WBRT — WBRT will be applied in 10 fractions with single doses of 3 Gy to the whole brain.
  Arms: Arm B: WBRT

SUMMARY:
Patients suffering from small cell lung cancer (SCLC) are at high risk for developing brain metastases (BM). To prevent a clinical manifestation of preexisting microscopic brain dissemination, prophylactic cranial irradiation (PCI) is offered to both limited and extensive disease patients, if they respond to first line regime, thus being at risk or at chance to develop clinical brain metastases. However, up to 10-15% of patients present with BM at initial diagnosis. If MRI is used as a diagnostic tool for initial staging the number even increases up to 15-20%. Additionally, between 40 - 50% of patients develop BM until time of death and the risk of developing BM further increases with prolonged survival. Treatment options are usually limited to WBRT and palliative chemotherapy but the actual effect of therapeutic WBRT has mainly been studied in small retrospective and nonrandomized studies. WBRT has been established as the treatment standard in patients with cerebral metastases from SCLC, however, it has only modest efficacy. Results might be improved by additional dose escalation. A SRS to cerebral metastases may be indicated in patients with intracranial disease, and the current protocol is aimed at exploring the neurocognition and efficacy of SCLC in patients with brain metastases treated with SRS or WBRT.

The present trial aims to exploratory investigate the treatment response to ´conventional whole brain radiotherapy´ (WBRT) and ´stereotactic radiotherapy´(SRS) in SCLC patients.

DETAILED DESCRIPTION:
Scientific Background: Patients suffering from BM from SCLC have a poor prognosis with a median survival ranging between 2-14 months. Treatment options for BM in SCLC are usually limited to WBRT, steroids or palliative chemotherapy. SCLC patients demonstrate an exception in the treatment of BM, because treatment options for a limited number of BM from other solid tumors commonly include surgery or SRS with or without WBRT. Even though SCLC is a radiosensitive tumor, higher doses are commonly not applied. Locally ablative treatments like SRS or surgery are less frequently used in patients with BM from SCLC as compared to other types of cancer due to the high incidence of brain metastases in SCLC and the increased likelihood of a diffuse failure pattern. It is of general belief that BM from SCLC are rarely solitary and usually occur at multiple sites. The investigators could not confirm these findings from this analysis as they found 1-5 BM in 39 % of their patients. WBRT, with a treatment time of about two weeks, is commonly the technique of choice for SCLC patients with any number of BM. In a recent Japanese trial, prophylactic cranial irradiation did not result in longer overall survival compared with observation in patients with early disease (ED) SCLC. PCI is therefore no longer recommended for patients with ED SCLC when patients receive regularly MRI examinations during follow-up.

Though, the initial response to cranial irradiation is good, especially in the synchronous setting, SCLC patients are at high risk of developing intracranial recurrence. In the investigators´ retrospective analysis median Overall survival (OS) after re-WBRT was only 2 months and the median OS after SRS was 6 months. These results are similar as compared to results for re-irradiation after PCI. In a recent analysis the investigators reported a prolonged survival for patients treated with SRS in the recurrent setting after previous PCI with a median survival of 5 months.

Therefore, the number of patients with oligometastatic cerebral disease might rise. Based on recursive partitioning Analysis (RPA) classification, the investigators found a median survival after WBRT of 17 months in RPA class I, 7 months in class II and 3 months in class III (p<0.0001), which is comparable to previous analyses using graded prognostic assessment (GPA) scoring. This is further of special interest as patients in RPA class I had a comparable or even better outcome than patients with non-cerebral disease treated with PCI. On the other hand, patients with RPA class III should be carefully selected for WBRT and treatment should be weighed against supportive therapy with steroids alone. This implicates that patient selection is mandatory, even in SCLC, and that the general paradigm of WBRT needs to be reevaluated.

Trial Objectives: The purpose of this trial is to explore the neurocognitive response in patients with brain metastases from SCLC treated with WBRT or SRS. The investigators proposed that patients treated with SRS would have inferior neurocognitive function based on the Hopkins Verbal Learning Test-Revised (HVLT-R) compared with patients treated with SRS alone.

Patients Selection: Patients with a diagnosis of brain metastases from SCLC will be evaluated and screened based on the protocol. All patients fulfilling the inclusion and exclusion criteria will be informed about the possibility to participate in the study. Registration for the study must be performed prior to beginning of RT. 56 patients will be enrolled in this exploratory clinical trial.

Trial Design: This pilot trial will be conducted as a single-center prospective, randomized, two-arm Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed small cell lung cancer (SCLC)
* Magentic resonance (MR)-imaging confirmed cerebral metastases (no resection, max. number of 10)
* age ≥ 18 years of Age
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

refusal of the patients to take part in the study

* previous radiotherapy of the brain
* Patients who have not yet recovered from acute high-grade toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another competing clinical study or observation period of competing trials, respectively
* MRI contraindication (i.e. cardiac pacemaker, implanted defibrillator, certain cardiac valve replacements, certain metal implants)
* Karnofsky score (KPS) <60
* Simultaneous cytotoxic chemotherapy
* Last application of chemotherapy/immunotherapy/targeted therapy <1 week before cerebral radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Neurocognition | 3 month after treatment
  Drop of at least 5 Points from baseline in HVLT-R test (Hopkins Verbal Learning Test-Revised)

SECONDARY OUTCOMES:
Intracranial progression | up to 12 month after treatment
  number of new cerebral metastases
Intracranial progression | up to 12 month after treatment
  Change in tumor size
Overall survival (OS) | 12 month OS
  Duration of survival defined as the interval between the date of RT begin and the date of death or date of leaving the study e.g., lost to follow up) whatever occurs first.
Death due to brain metastases | up to 12 month after treatment
  Death which directly connects to existing brain metastases
Locally progression-free survival | up to 12 month after treatment
  12 month Progression-fee survival referring to local tumour progression
Progression-free survival (PFS) | 12 month PFS
  12 month Progression-free survival
Changes in other cognitive performance measures | up to 12 month after treatment
  HVLT_R
Quality of life | up to 12 month after treatment
  BN20 QoL Questionaire
Quality of life | up to 12 month after treatment
  EORTC QoL Questionaire PAL (palliative)
Changes in other cognitive performance measures | up to 12 month after treatment
  CANTAB Test

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rieken, PD.Dr., Principal Investigator — chief senior physician in the department of Radiation Oncology
Locations (1):
- University Hospital of Heidelberg, Department of Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Auperin A, Arriagada R, Pignon JP, Le Pechoux C, Gregor A, Stephens RJ, Kristjansen PE, Johnson BE, Ueoka H, Wagner H, Aisner J. Prophylactic cranial irradiation for patients with small-cell lung cancer in complete remission. Prophylactic Cranial Irradiation Overview Collaborative Group. N Engl J Med. 1999 Aug 12;341(7):476-84. doi: 10.1056/NEJM199908123410703. PMID 10441603
- [Background] Bentzen SM, Constine LS, Deasy JO, Eisbruch A, Jackson A, Marks LB, Ten Haken RK, Yorke ED. Quantitative Analyses of Normal Tissue Effects in the Clinic (QUANTEC): an introduction to the scientific issues. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S3-9. doi: 10.1016/j.ijrobp.2009.09.040. PMID 20171515
- [Background] Bergqvist M, Brattstrom D, Bennmarker H, Wagenius G, Riska H, Brodin O. Irradiation of brain metastases from lung cancer: a retrospective study. Lung Cancer. 1998 Apr;20(1):57-63. doi: 10.1016/s0169-5002(98)00015-4. PMID 9699188
- [Background] Bernhardt D, Adeberg S, Bozorgmehr F, Opfermann N, Hoerner-Rieber J, Repka MC, Kappes J, Thomas M, Bischoff H, Herth F, Heussel CP, Debus J, Steins M, Rieken S. Nine-year Experience: Prophylactic Cranial Irradiation in Extensive Disease Small-cell Lung Cancer. Clin Lung Cancer. 2017 Jul;18(4):e267-e271. doi: 10.1016/j.cllc.2016.11.012. Epub 2016 Dec 2. PMID 28027850
- [Background] Bernhardt D, Adeberg S, Bozorgmehr F, Opfermann N, Hoerner-Rieber J, Konig L, Kappes J, Thomas M, Herth F, Heussel CP, Warth A, Debus J, Steins M, Rieken S. Outcome and prognostic factors in patients with brain metastases from small-cell lung cancer treated with whole brain radiotherapy. J Neurooncol. 2017 Aug;134(1):205-212. doi: 10.1007/s11060-017-2510-0. Epub 2017 May 30. PMID 28560661
- [Background] Bernhardt D, Bozorgmehr F, Adeberg S, Opfermann N, von Eiff D, Rieber J, Kappes J, Foerster R, Konig L, Thomas M, Debus J, Steins M, Rieken S. Outcome in patients with small cell lung cancer re-irradiated for brain metastases after prior prophylactic cranial irradiation. Lung Cancer. 2016 Nov;101:76-81. doi: 10.1016/j.lungcan.2016.09.010. Epub 2016 Sep 14. PMID 27794411
- [Background] van Buuren S. Multiple imputation of discrete and continuous data by fully conditional specification. Stat Methods Med Res. 2007 Jun;16(3):219-42. doi: 10.1177/0962280206074463. PMID 17621469
- [Background] Carmichael J, Crane JM, Bunn PA, Glatstein E, Ihde DC. Results of therapeutic cranial irradiation in small cell lung cancer. Int J Radiat Oncol Biol Phys. 1988 Mar;14(3):455-9. doi: 10.1016/0360-3016(88)90260-x. PMID 2830211
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Fertil B, Malaise EP. Intrinsic radiosensitivity of human cell lines is correlated with radioresponsiveness of human tumors: analysis of 101 published survival curves. Int J Radiat Oncol Biol Phys. 1985 Sep;11(9):1699-707. doi: 10.1016/0360-3016(85)90223-8. PMID 4030437
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Giannone L, Johnson DH, Hande KR, Greco FA. Favorable prognosis of brain metastases in small cell lung cancer. Ann Intern Med. 1987 Mar;106(3):386-9. doi: 10.7326/0003-4819-106-3-386. PMID 3028222
- [Background] Herfarth KK, Izwekowa O, Thilmann C, Pirzkall A, Delorme S, Hofmann U, Schadendorf D, Zierhut D, Wannenmacher M, Debus J. Linac-based radiosurgery of cerebral melanoma metastases. Analysis of 122 metastases treated in 64 patients. Strahlenther Onkol. 2003 Jun;179(6):366-71. doi: 10.1007/s00066-003-1050-z. PMID 12789461
- [Background] Hochstenbag MM, Twijnstra A, Wilmink JT, Wouters EF, ten Velde GP. Asymptomatic brain metastases (BM) in small cell lung cancer (SCLC): MR-imaging is useful at initial diagnosis. J Neurooncol. 2000 Jul;48(3):243-8. doi: 10.1023/a:1006427407281. PMID 11100822
- [Background] Kochhar R, Frytak S, Shaw EG. Survival of patients with extensive small-cell lung cancer who have only brain metastases at initial diagnosis. Am J Clin Oncol. 1997 Apr;20(2):125-7. doi: 10.1097/00000421-199704000-00003. PMID 9124183
- [Background] Komaki R, Cox JD, Whitson W. Risk of brain metastasis from small cell carcinoma of the lung related to length of survival and prophylactic irradiation. Cancer Treat Rep. 1981 Sep-Oct;65(9-10):811-4. PMID 6268295
- [Background] Lassen U, Kristjansen PE, Hansen HH. Brain metastases in small-cell lung cancer. Ann Oncol. 1995 Nov;6(9):941-4. doi: 10.1093/oxfordjournals.annonc.a059363. No abstract available. PMID 8624299
- [Background] Marks LB, Yorke ED, Jackson A, Ten Haken RK, Constine LS, Eisbruch A, Bentzen SM, Nam J, Deasy JO. Use of normal tissue complication probability models in the clinic. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S10-9. doi: 10.1016/j.ijrobp.2009.07.1754. PMID 20171502
- [Background] Newman SJ, Hansen HH. Proceedings: Frequency, diagnosis, and treatment of brain metastases in 247 consecutive patients with bronchogenic carcinoma. Cancer. 1974 Feb;33(2):492-6. doi: 10.1002/1097-0142(197402)33:23.0.co;2-o. No abstract available. PMID 4812766
- [Background] Nugent JL, Bunn PA Jr, Matthews MJ, Ihde DC, Cohen MH, Gazdar A, Minna JD. CNS metastases in small cell bronchogenic carcinoma: increasing frequency and changing pattern with lengthening survival. Cancer. 1979 Nov;44(5):1885-93. doi: 10.1002/1097-0142(197911)44:53.0.co;2-f. No abstract available. PMID 227582
- [Background] Postmus PE. Brain Metastases From Small Cell Lung Cancer: Chemotherapy, Radiotherapy, or Both? Semin Radiat Oncol. 1995 Jan;5(1):69-73. doi: 10.1054/SRAO00500069. PMID 10717129
- [Background] Quan AL, Videtic GM, Suh JH. Brain metastases in small cell lung cancer. Oncology (Williston Park). 2004 Jul;18(8):961-72; discussion 974, 979-80, 987. PMID 15328892
- [Background] Scharp M, Hauswald H, Bischof M, Debus J, Combs SE. Re-irradiation in the treatment of patients with cerebral metastases of solid tumors: retrospective analysis. Radiat Oncol. 2014 Jan 3;9:4. doi: 10.1186/1748-717X-9-4. PMID 24387239
- [Background] Schwartz LH, Seymour L, Litiere S, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, de Vries E. RECIST 1.1 - Standardisation and disease-specific adaptations: Perspectives from the RECIST Working Group. Eur J Cancer. 2016 Jul;62:138-45. doi: 10.1016/j.ejca.2016.03.082. Epub 2016 May 26. PMID 27237360
- [Background] Schwer AL, Gaspar LE. Update in the treatment of brain metastases from lung cancer. Clin Lung Cancer. 2006 Nov;8(3):180-6. doi: 10.3816/CLC.2006.n.045. PMID 17239293
- [Background] Shibamoto Y, Baba F, Oda K, Hayashi S, Kokubo M, Ishihara S, Itoh Y, Ogino H, Koizumi M. Incidence of brain atrophy and decline in mini-mental state examination score after whole-brain radiotherapy in patients with brain metastases: a prospective study. Int J Radiat Oncol Biol Phys. 2008 Nov 15;72(4):1168-73. doi: 10.1016/j.ijrobp.2008.02.054. Epub 2008 May 19. PMID 18495375
- [Background] Slotman B, Faivre-Finn C, Kramer G, Rankin E, Snee M, Hatton M, Postmus P, Collette L, Musat E, Senan S; EORTC Radiation Oncology Group and Lung Cancer Group. Prophylactic cranial irradiation in extensive small-cell lung cancer. N Engl J Med. 2007 Aug 16;357(7):664-72. doi: 10.1056/NEJMoa071780. PMID 17699816
- [Background] Soffietti R, Kocher M, Abacioglu UM, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Mueller RP, Tridello G, Collette L, Bottomley A. A European Organisation for Research and Treatment of Cancer phase III trial of adjuvant whole-brain radiotherapy versus observation in patients with one to three brain metastases from solid tumors after surgical resection or radiosurgery: quality-of-life results. J Clin Oncol. 2013 Jan 1;31(1):65-72. doi: 10.1200/JCO.2011.41.0639. Epub 2012 Dec 3. PMID 23213105
- [Background] Son CH, Jimenez R, Niemierko A, Loeffler JS, Oh KS, Shih HA. Outcomes after whole brain reirradiation in patients with brain metastases. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):e167-72. doi: 10.1016/j.ijrobp.2011.03.020. Epub 2011 May 27. PMID 21620583
- [Background] Sperduto PW, Chao ST, Sneed PK, Luo X, Suh J, Roberge D, Bhatt A, Jensen AW, Brown PD, Shih H, Kirkpatrick J, Schwer A, Gaspar LE, Fiveash JB, Chiang V, Knisely J, Sperduto CM, Mehta M. Diagnosis-specific prognostic factors, indexes, and treatment outcomes for patients with newly diagnosed brain metastases: a multi-institutional analysis of 4,259 patients. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):655-61. doi: 10.1016/j.ijrobp.2009.08.025. Epub 2009 Nov 26. PMID 19942357
- [Background] Sperduto PW, Kased N, Roberge D, Xu Z, Shanley R, Luo X, Sneed PK, Chao ST, Weil RJ, Suh J, Bhatt A, Jensen AW, Brown PD, Shih HA, Kirkpatrick J, Gaspar LE, Fiveash JB, Chiang V, Knisely JP, Sperduto CM, Lin N, Mehta M. Summary report on the graded prognostic assessment: an accurate and facile diagnosis-specific tool to estimate survival for patients with brain metastases. J Clin Oncol. 2012 Feb 1;30(4):419-25. doi: 10.1200/JCO.2011.38.0527. Epub 2011 Dec 27. PMID 22203767
- [Background] Takahashi T, Yamanaka T, Seto T, Harada H, Nokihara H, Saka H, Nishio M, Kaneda H, Takayama K, Ishimoto O, Takeda K, Yoshioka H, Tachihara M, Sakai H, Goto K, Yamamoto N. Prophylactic cranial irradiation versus observation in patients with extensive-disease small-cell lung cancer: a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2017 May;18(5):663-671. doi: 10.1016/S1470-2045(17)30230-9. Epub 2017 Mar 23. PMID 28343976
- [Background] Tsao MN, Lloyd N, Wong RK, Chow E, Rakovitch E, Laperriere N, Xu W, Sahgal A. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD003869. doi: 10.1002/14651858.CD003869.pub3. PMID 22513917
- [Background] Welzel G, Fleckenstein K, Schaefer J, Hermann B, Kraus-Tiefenbacher U, Mai SK, Wenz F. Memory function before and after whole brain radiotherapy in patients with and without brain metastases. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1311-8. doi: 10.1016/j.ijrobp.2008.03.009. Epub 2008 Apr 28. PMID 18448270
- [Background] Wong WW, Schild SE, Sawyer TE, Shaw EG. Analysis of outcome in patients reirradiated for brain metastases. Int J Radiat Oncol Biol Phys. 1996 Feb 1;34(3):585-90. doi: 10.1016/0360-3016(95)02156-6. PMID 8621282
- [Derived] Bernhardt D, Hommertgen A, Schmitt D, El Shafie R, Paul A, Konig L, Mair-Walther J, Krisam J, Klose C, Welzel T, Horner-Rieber J, Kappes J, Thomas M, Heussel CP, Steins M, Kieser M, Debus J, Rieken S. Whole brain radiation therapy alone versus radiosurgery for patients with 1-10 brain metastases from small cell lung cancer (ENCEPHALON Trial): study protocol for a randomized controlled trial. Trials. 2018 Jul 16;19(1):388. doi: 10.1186/s13063-018-2745-x. PMID 30012190